CLINICAL TRIAL: NCT04219696
Title: Determining the Optimal Dose of Reactive Balance Training After Stroke - a Pilot Study
Brief Title: Determining the Optimal Dose of Reactive Balance Training After Stroke
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: Heart and Stroke Foundation Canadian Partnership for Stroke Recovery (Unknown)
Responsible Party: Principal Investigator, Avril Mansfield, Scientist, Toronto Rehabilitation Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-6001
Record Dates: First submitted 2019-12-17; First posted 2020-01-07 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome measures will be obtained by a research assistant who will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 session (Active Comparator): Participants will complete one 45-minute session of reactive balance training. Participants will experience 40-60 perturbations during this session. Participants will also complete 5 45-minute 'traditional' balance training sessions.
  Interventions: Other: Reactive balance training
- 3 sessions (Experimental): Participants will complete three 45-minute sessions of reactive balance training. Participants will experience 40-60 perturbations during each session. Participants will also complete 3 45-minute 'traditional' balance training sessions.
  Interventions: Other: Reactive balance training
- 6 sessions (Experimental): Participants will complete six 45-minute sessions of reactive balance training. Participants will experience 40-60 perturbations during each session.
  Interventions: Other: Reactive balance training

INTERVENTIONS:
Other: Reactive balance training — A research physiotherapist will oversee reactive balance training (RBT) to ensure consistent RBT delivery across participants. Training strategies will be individualized to each participant, based on their balance impairments and rehabilitation goals. The RBT program includes multi-directional 'internal' and 'external' balance perturbations. Internal perturbations are achieved by asking the participant to complete tasks that challenge balance control, such that they lose balance when attempting to perform the task (e.g., kicking a soccer ball). External perturbation are delivered manually using a push or pull from the physiotherapist. As participants improve their reactive balance control, difficulty will be increased by shifting task requirements along a continuum from stable to mobile, and from predictable to unpredictable, and by increasing perturbation magnitude or imposing sensory or environmental challenges.

SUMMARY:
Falls in daily life are one of the most significant complications for people with stroke. Fall rates are particularly high soon after discharge from stroke rehabilitation. A new type of balance training, called reactive balance training (RBT), can reduce fall rates after discharge from stroke rehabilitation. In our previous study, RBT was implemented as part of routine care, and as a result, the dose of training was different for each participant; participants completed between one and twelve 30-minute sessions of RBT. Previous research in healthy older adults suggests that a single session of RBT is enough to lead to lasting changes in reactive balance control and reduce fall rates in daily life. It is not clear if the same is true for people with stroke, who have more severe impairments and might need a higher dose of training to achieve the same benefits.

The overall goal of this work is to determine the optimal dose of reactive balance training for people with stroke who are attending rehabilitation. This pilot study will determine the feasibility of a clinical trial to address this larger goal. People with sub-acute stroke will be randomly assigned to one of three groups: 1 session, 3 sessions, or 6 sessions of RBT. Each session will be 45 minutes long, and will occur as part of participants' routine out-patient rehabilitation. We will use our experiences with this pilot study to help design a larger study. Specifically, we will use this pilot study to answer the following questions: 1) what is the optimal sample size; 2) how long will it take to reach this sample size; 3) what outcome measures should be used; 4) how feasible is it to prescribe a specific dose of RBT to people with sub-acute stroke; and 5) what two intervention groups should be included in the larger trial?

ELIGIBILITY:
Inclusion criteria:

* Sub-acute stroke;
* Receiving out-patient rehabilitation at the Toronto Rehabilitation Institute;
* Can stand independently for >30 seconds;
* Can walk with or without a gait aid (but without assistance of another person) for >10 metres; and
* Living in the community.

Exclusion Criteria:

* Completed reactive balance training during in-patient rehabilitation;
* Lower-extremity amputation, weight-bearing restrictions, recent lower-extremity injury or surgery (e.g., fracture), acute back or lower-limb pain, halo, aspen collar, history of fragility fracture and/or severe osteoporosis/osteopenia, contractures that prevent neutral hip or ankle;
* Activity restrictions following cardiac event/surgery, abnormal or unstable cardiovascular responses to exercise, arterial dissection;
* Severe spasticity in the legs;
* Cognitive impairment (i.e., unable to understand the purpose of training and/or to provide informed consent); and/or
* Acute illness (e.g., vomiting, fever), extreme obesity (exceeds safety harness weight limits), colostomy bags, indwelling catheter, infection, pressure sore on pelvis or trunk.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Rate of falls in daily life | 6 months post-discharge
  Participants will be asked to report falls ("an event that results in a person coming to rest unintentionally on the ground or other lower level") in the 6 months post-training. Participants will be provided with stamped, addressed postcards to mail to the research team every 2 weeks for 6 months post-training. Postcards will contain a calendar, on which participants will record falls. The research assistant will call participants who do not return the postcard to determine if any falls occurred. The research assistant will contact participants reporting a fall to complete a short questionnaire determining the cause and consequences of the fall.

SECONDARY OUTCOMES:
Rate of accrual | Through study completion, an average of 18 months
  Number of participants recruited per month
Rate of missing data | Through study completion, an average of 18 months
  Number of complete datasets for each of the other pre-specified outcomes
Compliance with the intervention | Through study completion, an average of 18 months
  Number of prescribed training sessions attended

OTHER OUTCOMES:
Chedoke-McMaster Stroke Assessment | Pre-intervention (at admission), post-intervention (before discharge, approximately 4 weeks), and 6 months post-intervention
  Construct: motor recovery. Range: 1-7. Higher scores indicate improved recovery.
Mini-Balance Evaluation Systems Test | Pre-intervention (at admission), post-intervention (before discharge, approximately 4 weeks), and 6 months post-intervention
  Construct: Anticipatory balance control, reactive balance control, gait, and sensory orientation in balance. Scale range: 0-28 (total), 0-6 (anticipatory balance control), 0-6 (reactive balance control), 0-10 (gait), 0-6 (sensory orientation). Higher values represent improved outcome. The total score is created by adding the sub-scale scores
Activities-specific Balance Confidence Scale | Pre-intervention (at admission), post-intervention (before discharge, approximately 4 weeks), and 6 months post-intervention
  Construct: balance confidence. Scale range: 0-100. Higher values represent improved outcome
Reactive balance control following novel unpredictable postural perturbation | Pre-intervention (at admission), post-intervention (before discharge, approximately 4 weeks), and 6 months post-intervention
  Participants will be outfitted with reflective markers, and will complete 8-10 walking trials on a movable platform. On one trial, the platform will move forward suddenly on heel strike to trigger a slip-like perturbation. On another trial, the platform will move backward suddenly on toe-off to trigger a trip-like perturbation. The platform will only move during these two trials, such that the perturbation will be unpredictable to participants. These perturbations differ from what will be used during training, and will measure transfer of training to novel and ecological loss of balance. Biomechanical stability when responding to the perturbation will be measured using an established method that considers the distance between the centre of mass and base of support; in general, a more posteriorly- (slip) or anteriorly-located (trip) centre of mass is considered less stable.
Physical Activity Scale for Individuals with Physical Disabilities | Average of three scores at approximately 2-, 4- and 6-months post-discharge
  Construct: physical activity in daily life. Scale range: not applicable (the maximum score that is technically achievable would not be feasible). Higher scores represent improved outcome
Subjective Index of Physical and Social Outcome | Average of three scores at approximately 2-, 4- and 6-months post-discharge
  Construct: participation Scale range: 0-40 (total); 0-20 (social sub-scale), 0-20 (physical sub-scale). Higher scores represent improved outcome. The total score is the sum of the sub-scale scores

CONTACTS AND LOCATIONS:
Overall Officials: Avril Mansfield, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Rehabilitation Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mansfield A, Inness EL, Danells CJ, Jagroop D, Bhatt T, Huntley AH. Determining the optimal dose of reactive balance training after stroke: study protocol for a pilot randomised controlled trial. BMJ Open. 2020 Aug 26;10(8):e038073. doi: 10.1136/bmjopen-2020-038073. PMID 32847916